CLINICAL TRIAL: NCT01088542
Title: The Interplay of Social, Normative, and Legal Marijuana Environments and Marijuana and ATOD Use From Late Childhood to Young Adulthood
Brief Title: The Community Youth Development Study: A Test of Communities That Care
Acronym: CYDS IV
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Margaret Kuklinski, Senior Research Scientist, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00000692; R01DA044522 (NIH)
Record Dates: First submitted 2010-03-15; First posted 2010-03-17 (Estimated); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Substance Abuse; Juvenile Delinquency; Sexual Behavior; Criminal Behavior; Violence; Depression; Anxiety; Suicide; Sexually Transmitted Infection; Educational Attainment
Keywords: substance use; delinquency; risky sexual behavior; risk factors; protective factors; prevention; community coalitions; systems transformation; violence
MeSH Terms: conditions — Substance-Related Disorders; Sexual Behavior; Criminal Behavior; Depression; Anxiety Disorders; Suicide; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No intervention (No Intervention): Communities in the no intervention arm received no intervention from the project and continued to implement prevention services as usual.
- Communities That Care Intervention (Experimental): Communities randomly assigned to the experimental condition received 5 years of training and technical assistance (from 2003 to 2008) to implement the Communities That Care (CTC) prevention system in their communities. They also received 5 years of funding to support a full-time community coordinator and 4 years of seed money to implement tested and effective prevention programs selected as a result of their CTC process.
  Interventions: Behavioral: Communities That Care

INTERVENTIONS:
Behavioral: Communities That Care — The Communities That Care (CTC) system provides communities training and ongoing technical assistance in a structured process for conducting prevention needs assessments using epidemiological data on levels of risk and protective factors for adolescent problem behaviors, selection of tested and effective preventive interventions shown to address community-prioritized factors, implementation of these interventions with fidelity, and evaluation of the community's progress toward its goals. The CTC system is designed to produce a plan for prevention services that is tailored to the needs of each community. CTC is installed in five phases through a manualized series of training events designed to build the capacity of communities to install and sustain the system over time.
  Arms: Communities That Care Intervention

SUMMARY:
The Community Youth Development Study is an experimental test of the Communities That Care (CTC) prevention planning system. It has been designed to find out if communities that were trained to use the CTC system improved public health by reducing rates of adolescent drug use, delinquency, violence, and risky sexual behavior when compared to communities that did not use this approach. The primary purpose of the current continuation study is to investigate whether CTC has long-term effects on substance use, antisocial behavior, and violence, as well as secondary effects on educational attainment, mental health, and sexual risk behavior in young adults at ages 26 and 28. The continuation study also examines (a) how the interaction of social, normative, and legal marijuana contexts creates variation in the permissiveness of individuals' marijuana environments from late childhood to young adulthood and (b) whether, when, and for whom permissive marijuana environments increase marijuana and ATOD use and misuse from age 11 to 28 and interfere with the adoption of adult roles.

DETAILED DESCRIPTION:
Preventing alcohol, tobacco, and other drug use; delinquency; violence; and health-risking sexual behavior among adolescents is a national priority. While advances in prevention science over the past two decades have produced a growing list of tested and effective programs and policies for preventing these behaviors, widespread dissemination and high-quality implementation of these effective programs and policies in communities has not been achieved. The development and testing of approaches for translating prevention research findings into effective community prevention service systems with long-term impact is important to achieving reductions in the prevalence of adolescent health and behavior problems that are sustained into adulthood.

The Community Youth Development Study (CYDS) is a community-randomized trial of the effects of Communities That Care (CTC) on community prevention systems and adolescent risk, protection, and behavioral health outcomes. The current continuation study is evaluating the long-term effects of CTC on a panel of 4,407 young adults at ages 21 and 23 who have been surveyed regularly since the trial started when they were in grade 5.

CTC is a prevention planning and capacity building system for improving behavioral health problems among youth community-wide. CTC guides communities to implement with fidelity and monitor the results of effective prevention programs that address community-specific elevated risk factors and depressed protective factors and reduce problem behavior. The CTC system is hypothesized first to produce improvements in key characteristics of community prevention service systems, which, in turn, reduce community levels of risk, increase protective factors, and lower rates of youth problem behaviors.

The CYDS communities were matched in pairs within state, on population size, racial and ethnic diversity, economic indicators, and crime rates. One community from each matched pair was assigned randomly by a coin toss to either the intervention or control condition. Starting in 2003, intervention communities received training, technical assistance, and materials and funding needed to install the CTC prevention system in years 2-5 (2004-2008), hire a community coordinator, and implement 2-5 tested preventive interventions. Selected interventions addressed local prevention priorities established by communities after reviewing local epidemiological data on youth risk factors, protective factors and problem behaviors. Control communities received no training or technical assistance from the study. Technical assistance and study-provided funding to intervention communities ended after 5 years.

The initial CYDS trial (2003-2008) evaluated the efficacy of CTC in reducing levels of risk, increasing levels of protection, and reducing levels of drug use and other problem behaviors in adolescents from Grades 5 through 9. It also tested the effects of CTC on prevention service system transformation (e.g., increases in a science-based approach to prevention, collaboration among prevention service organizations, support for prevention, community norms against drug use and delinquency, and use of the Social Development Strategy to guide interactions with youth) as reported by key community leaders and members of CTC coalitions.

The first continuation study (2009-2013) assessed the effects of installation and implementation of CTC when panel youth were in Grades 10 through Age 19. During this period, panel youth passed through high school, the developmental period of greatest risk for delinquent and violent behavior, and a period of greatly increasing substance use and problems related to substance use. The study evaluated the long-term effects of CTC on adolescent and young adult risk and problem behaviors, including primary outcomes of substance use and abuse, delinquency, crime, and violence. It also evaluated the sustainability of the CTC prevention system without the study-provided funding and support that were offered during the implementation of CTC in the 12 intervention communities during the initial efficacy trial.

The second continuation study (2013-2017) investigated the long-term effects of CTC on young adult substance use and misuse, crime, violence, and incarceration 11 and 13 years following CTC's initial installation. It also evaluated possible effects on a number of secondary outcomes salient in young adulthood, including HIV/AIDS sexual risk behavior, depression and suicidality, anxiety and other mental health disorders, and educational attainment. Panel youth were surveyed twice during the study, at ages 21 and 23.

The third continuation study (2018-2023) further investigates the long-term effects of CTC on the study's primary outcomes of substance use and misuse, crime, violence, and incarceration 16 and 18 years after CTC was installed in intervention communities. As in the prior continuation, it will also evaluate possible long-term effects on salient secondary outcomes, including HIV/AIDS sexual risk behavior, depression and suicidality, anxiety and other mental health disorders, and educational attainment. Another major aim of this study is to examine the normative and legal environment around marijuana use in the U.S., which is becoming more permissive, raising concern that it will increase youth and young adult marijuana and other drug use and associated negative consequences including addiction. Understanding how marijuana use norms and behaviors in multiple social contexts (e.g., peer, family, and community) interact with the legal marijuana context and impact drug use behavior from age 11 to 28 will assist in the identification of malleable targets for interventions and public health approaches to prevent the possible negative outcomes of increasing permissiveness towards marijuana use. Panel participants will be surveyed twice, at ages 26 and 28.

ELIGIBILITY:
Inclusion Criteria:

* Resident at baseline in one of the 24 participating communities
* Student in the Class of 2011 panel sample or in grades 6, 8, 10, or 12 during a survey year
* Community leader or prevention service provider in one of the participating communities

Exclusion Criteria:

* Unable to read and comprehend consent materials and/or survey questions in either english or spanish

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52323 (Actual)
Dates: Start 2003-10-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Targeted risk and protective factors, substance use, delinquency, violence | Baseline through thirteen-year follow-up (age 23)
  Surveys of the panel starting in 5th grade (2004) and continuing in grades 6-10, grade 12, and at ages 19, 21, and 23 are used to assess the impact of the intervention on risk and protective factors targeted by communities, substance use, delinquency, and violence. Cross-sectional surveys of all youth in grades 6, 8, 10, and 12 in all participating communities, conducted every 2 years from 2002 through 2012, are also used to assess the impact of the intervention on these primary outcomes.
CTC coalition functioning, prevention system transformation, evidence-based program (EBP) implementation | Baseline through eight-year follow-up (age 18)
  Structured telephone interviews with key community leaders, CTC coalition members, and prevention services providers (Community Key Informant Survey, Coalition Board Interview, Community Resource Documentation Survey) conducted in 2001-02, 2004-05, 2007-08, 2009-10, and 2011-12 are used to assess intervention effects on CTC coalition functioning, prevention system transformation, and evidence-based prevention program implementation.

SECONDARY OUTCOMES:
Substance use disorder, depression and generalized anxiety disorder, sexual risk behavior | Nine- through thirteen-year follow-up
  Secondary outcomes salient in late adolescence and young adulthood were added to the self-report longitudinal survey beginning at the nine-year follow-up (age 19).

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Kuklinski, Ph.D., Principal Investigator — University of Washington; Sabrina Oesterle, Ph.D., Principal Investigator — University of Arizona
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
We support the goal of making datasets available to researchers in a timely manner to expedite translation of research results into knowledge, products, and procedures to improve human health. With these goals in mind, we have entered into data-sharing collaborations many times with outside researchers. To ensure that the use of these data stay within the legal and ethical constraints of the consent agreement under which they were collected, we have developed a Fair Use Agreement, available upon request, that is signed by the Principal Investigator, Dr. Kuklinski, and by the collaborating researcher when agreement has been reached to share study data. As part of the Fair Use Agreement, we ask researchers to abide by the same Data and Safety Monitoring Plan (DSMP) that we adhere to. We will continue to share data with other researchers who meet the terms of our Fair Use Agreement (and DSMP) and share our strong commitment to protection of the rights and privacy of study participants.

REFERENCES:
- [Background] Oesterle S, Kuklinski MR, Hawkins JD, Skinner ML, Guttmannova K, Rhew IC. Long-Term Effects of the Communities That Care Trial on Substance Use, Antisocial Behavior, and Violence Through Age 21 Years. Am J Public Health. 2018 May;108(5):659-665. doi: 10.2105/AJPH.2018.304320. Epub 2018 Mar 22. PMID 29565666
- [Background] Rhew IC, Oesterle S, Coffman D, Hawkins JD. Effects of Exposure to the Communities That Care Prevention System on Youth Problem Behaviors in a Community-Randomized Trial: Employing an Inverse Probability Weighting Approach. Eval Health Prof. 2018 Jun;41(2):270-289. doi: 10.1177/0163278718759397. Epub 2018 Feb 20. PMID 29463119
- [Background] Oesterle S, Hawkins JD, Kuklinski MR, Fagan AA, Fleming C, Rhew IC, Brown EC, Abbott RD, Catalano RF. Effects of Communities That Care on Males' and Females' Drug Use and Delinquency 9 Years After Baseline in a Community-Randomized Trial. Am J Community Psychol. 2015 Dec;56(3-4):217-28. doi: 10.1007/s10464-015-9749-4. PMID 26377418
- [Result] Rhew IC, Hawkins JD, Murray DM, Fagan AA, Oesterle S, Abbott RD, Catalano RF. Evaluation of Community-Level Effects of Communities That Care on Adolescent Drug Use and Delinquency Using a Repeated Cross-Sectional Design. Prev Sci. 2016 Feb;17(2):177-87. doi: 10.1007/s11121-015-0613-4. PMID 26462492
- [Result] Gloppen KM, Brown EC, Wagenaar BH, Hawkins JD, Rhew IC, Oesterle S. Sustaining Adoption of Science-based Prevention Through Communities That Care. J Community Psychol. 2016 Jan;44(1):78-89. doi: 10.1002/jcop.21743. Epub 2015 Dec 18. No abstract available. PMID 27397946
- [Result] Kim BK, Gloppen KM, Rhew IC, Oesterle S, Hawkins JD. Effects of the communities that care prevention system on youth reports of protective factors. Prev Sci. 2015 Jul;16(5):652-62. doi: 10.1007/s11121-014-0524-9. PMID 25366931
- [Result] Kim BK, Oesterle S, Hawkins JD, Shapiro VB. Assessing Sustained Effects of Communities That Care on Youth Protective Factors. J Soc Social Work Res. 2015 Winter;6(4):565-589. doi: 10.1086/684163. Epub 2015 Oct 6. PMID 26951879
- [Result] Kuklinski MR, Fagan AA, Hawkins JD, Briney JS, Catalano RF. Benefit-Cost Analysis of a Randomized Evaluation of Communities That Care: Monetizing Intervention Effects on the Initiation of Delinquency and Substance Use Through Grade 12. J Exp Criminol. 2015 Jun 1;11(2):165-192. doi: 10.1007/s11292-014-9226-3. PMID 26213527
- [Result] Shapiro VB, Hawkins JD, Oesterle S. Building Local Infrastructure for Community Adoption of Science-Based Prevention: The Role of Coalition Functioning. Prev Sci. 2015 Nov;16(8):1136-46. doi: 10.1007/s11121-015-0562-y. PMID 26017632
- [Result] Shapiro VB, Oesterle S, Hawkins JD. Relating coalition capacity to the adoption of science-based prevention in communities: evidence from a randomized trial of Communities That Care. Am J Community Psychol. 2015 Mar;55(1-2):1-12. doi: 10.1007/s10464-014-9684-9. PMID 25323784
- [Result] Brown EC, Hawkins JD, Rhew IC, Shapiro VB, Abbott RD, Oesterle S, Arthur MW, Briney JS, Catalano RF. Prevention system mediation of communities that care effects on youth outcomes. Prev Sci. 2014 Oct;15(5):623-32. doi: 10.1007/s11121-013-0413-7. PMID 23828448
- [Result] Hawkins JD, Oesterle S, Brown EC, Abbott RD, Catalano RF. Youth problem behaviors 8 years after implementing the communities that care prevention system: a community-randomized trial. JAMA Pediatr. 2014 Feb;168(2):122-9. doi: 10.1001/jamapediatrics.2013.4009. PMID 24322060
- [Result] Oesterle S, Hawkins JD, Fagan AA, Abbott RD, Catalano RF. Variation in the sustained effects of the communities that care prevention system on adolescent smoking, delinquency, and violence. Prev Sci. 2014 Apr;15(2):138-145. doi: 10.1007/s11121-013-0365-y. PMID 23412948
- [Result] Kuklinski MR, Hawkins JD, Plotnick RD, Abbott RD, Reid CK. How has the economic downturn affected communities and implementation of science-based prevention in the randomized trial of communities that care? Am J Community Psychol. 2013 Jun;51(3-4):370-84. doi: 10.1007/s10464-012-9557-z. PMID 23054169
- [Result] Monahan KC, Hawkins JD, Abbott RD. The application of meta-analysis within a matched-pair randomized control trial: an illustration testing the effects of communities that care on delinquent behavior. Prev Sci. 2013 Feb;14(1):1-12. doi: 10.1007/s11121-012-0298-x. PMID 23111547
- [Result] Rhew IC, Brown EC, Hawkins JD, Briney JS. Sustained effects of the Communities That Care system on prevention service system transformation. Am J Public Health. 2013 Mar;103(3):529-35. doi: 10.2105/AJPH.2011.300567. Epub 2012 Jun 21. PMID 22720764
- [Result] Shapiro VB, Hawkins JD, Oesterle S, Monahan KC, Brown EC, Arthur MW. Variation in the Effect of Communities That Care on Community Adoption of a Scientific Approach to Prevention. J Soc Social Work Res. 2013 Aug 20;4(3):10.5243/jsswr.2013.10. doi: 10.5243/jsswr.2013.10. PMID 24319545
- [Result] Steketee M, Oesterle S, Jonkman H, Hawkins JD, Haggerty KP, Aussems C. Transforming prevention systems in the United States and the Netherlands using Communities That Care Promising prevention in the eyes of Josine Junger-Tas. Eur J Crim Pol Res. 2013 Jun 1;19(2):99-116. doi: 10.1007/s10610-012-9194-y. PMID 24465089
- [Result] Fagan AA, Hanson K, Briney JS, David Hawkins J. Sustaining the utilization and high quality implementation of tested and effective prevention programs using the communities that care prevention system. Am J Community Psychol. 2012 Jun;49(3-4):365-77. doi: 10.1007/s10464-011-9463-9. PMID 21809149
- [Result] Gloppen KM, Arthur MW, Hawkins JD, Shapiro VB. Sustainability of the Communities That Care prevention system by coalitions participating in the Community Youth Development Study. J Adolesc Health. 2012 Sep;51(3):259-64. doi: 10.1016/j.jadohealth.2011.12.018. Epub 2012 Mar 3. PMID 22921136
- [Result] Hawkins JD, Oesterle S, Brown EC, Monahan KC, Abbott RD, Arthur MW, Catalano RF. Sustained decreases in risk exposure and youth problem behaviors after installation of the Communities That Care prevention system in a randomized trial. Arch Pediatr Adolesc Med. 2012 Feb;166(2):141-8. doi: 10.1001/archpediatrics.2011.183. Epub 2011 Oct 3. PMID 21969362
- [Result] Kuklinski MR, Briney JS, Hawkins JD, Catalano RF. Cost-benefit analysis of communities that care outcomes at eighth grade. Prev Sci. 2012 Apr;13(2):150-61. doi: 10.1007/s11121-011-0259-9. PMID 22108900
- [Result] Brown EC, Hawkins JD, Arthur MW, Briney JS, Fagan AA. Prevention Service System Transformation Using Communities That Care. J Community Psychol. 2011 Mar 1;39(2):183-201. doi: 10.1002/jcop.20426. PMID 23606774
- [Result] Fagan AA, Arthur MW, Hanson K, Briney JS, Hawkins JD. Effects of Communities That Care on the adoption and implementation fidelity of evidence-based prevention programs in communities: results from a randomized controlled trial. Prev Sci. 2011 Sep;12(3):223-34. doi: 10.1007/s11121-011-0226-5. PMID 21667142
- [Result] Arthur MW, Hawkins JD, Brown EC, Briney JS, Oesterle S; Social Development Research Group; Abbott RD. Implementation of the Communities That Care Prevention System by Coalitions in the Community Youth Development Study. J Community Psychol. 2010 Mar;38(2):245-258. doi: 10.1002/jcop.20362. PMID 22199409
- [Result] Oesterle S, Hawkins JD, Fagan AA, Abbott RD, Catalano RF. Testing the universality of the effects of the communities that care prevention system for preventing adolescent drug use and delinquency. Prev Sci. 2010 Dec;11(4):411-23. doi: 10.1007/s11121-010-0178-1. PMID 20422289
- [Result] Brown EC, Graham JW, Hawkins JD, Arthur MW, Baldwin MM, Oesterle S, Briney JS, Catalano RF, Abbott RD. Design and analysis of the Community Youth Development Study longitudinal cohort sample. Eval Rev. 2009 Aug;33(4):311-34. doi: 10.1177/0193841X09337356. Epub 2009 Jun 9. PMID 19509119
- [Result] Fagan AA, Hanson K, Hawkins JD, Arthur M. Translational Research in Action: Implementation of the Communities That Care Prevention System in 12 Communities. J Community Psychol. 2009 Sep;37(7):809-829. doi: 10.1002/jcop.20332. PMID 22121303
- [Result] Hawkins JD, Oesterle S, Brown EC, Arthur MW, Abbott RD, Fagan AA, Catalano RF. Results of a type 2 translational research trial to prevent adolescent drug use and delinquency: a test of Communities That Care. Arch Pediatr Adolesc Med. 2009 Sep;163(9):789-98. doi: 10.1001/archpediatrics.2009.141. PMID 19736331
- [Result] Fagan AA, Hanson K, Hawkins JD, Arthur MW. Implementing effective community-based prevention programs in the Community Youth Development Study. Youth Violence and Juvenile Justice 6(3):256-278, 2008.
- [Result] Fagan AA, Hanson K, Hawkins JD, Arthur MW. Bridging science to practice: achieving prevention program implementation fidelity in the community youth development study. Am J Community Psychol. 2008 Jun;41(3-4):235-49. doi: 10.1007/s10464-008-9176-x. PMID 18302016
- [Result] Hawkins JD, Brown EC, Oesterle S, Arthur MW, Abbott RD, Catalano RF. Early effects of Communities That Care on targeted risks and initiation of delinquent behavior and substance use. J Adolesc Health. 2008 Jul;43(1):15-22. doi: 10.1016/j.jadohealth.2008.01.022. Epub 2008 Apr 18. PMID 18565433
- [Result] Hawkins JD, Catalano RF, Arthur MW, Egan E, Brown EC, Abbott RD, Murray DM. Testing communities that care: the rationale, design and behavioral baseline equivalence of the community youth development study. Prev Sci. 2008 Sep;9(3):178-90. doi: 10.1007/s11121-008-0092-y. Epub 2008 May 31. PMID 18516681
- [Result] Quinby RK, Fagan AA, Hanson K, Brooke-Weiss B, Arthur MW, Hawkins JD. Installing the Communities That Care prevention system: Implementation progress and fidelity in a randomized controlled trial. Journal of Community Psychology 36(3):313-332, 2008.
- [Result] Brown EC, Hawkins JD, Arthur MW, Briney JS, Abbott RD. Effects of Communities That Care on prevention services systems: findings from the community youth development study at 1.5 years. Prev Sci. 2007 Sep;8(3):180-91. doi: 10.1007/s11121-007-0068-3. Epub 2007 Jun 30. PMID 17602298
- [Result] Van Horn ML, Fagan AA, Hawkins JD, Oesterle S. Effects of the Communities That Care system on cross-sectional profiles of adolescent substance use and delinquency. Am J Prev Med. 2014 Aug;47(2):188-97. doi: 10.1016/j.amepre.2014.04.004. Epub 2014 Jun 27. PMID 24986217
- [Derived] Kuklinski MR, Gibbons BJ, Bowser DM, McCollister KE, Smart R, Dunlap LJ, Shenkar E, Bonar EE, Boomer T, Campbell M, Fiellin LE, Hutton DW, Rao V, Saldana L, Su K, Walton MA, Yilmazer T. Investing in Interventions to Prevent Opioid Use Disorder in Adolescents and Young Adults: Start-up Costs from NIDA's HEAL Prevention Initiative. Prev Sci. 2025 Nov;26(7):1045-1055. doi: 10.1007/s11121-025-01835-6. Epub 2025 Oct 14. PMID 41085955
- [Derived] Rowhani-Rahbar A, Oesterle S, Gause EL, Kuklinski MR, Ellyson AM, Schleimer JP, Dalve K, Weybright EH, Briney JS, Hawkins JD. Effect of the Communities That Care Prevention System on Adolescent Handgun Carrying: A Cluster-Randomized Clinical Trial. JAMA Netw Open. 2023 Apr 3;6(4):e236699. doi: 10.1001/jamanetworkopen.2023.6699. PMID 37022682
- [Derived] Guttmannova K, Oesterle S, Skinner ML, Kuklinski MR, Hultgren B, Rhew IC, Parker M, Briney JS, White HR. Substance-Specific Risk Factors among Young Adults: Potential Prevention Targets across Cannabis-Permissive Environments. Subst Use Misuse. 2022;57(13):1923-1930. doi: 10.1080/10826084.2022.2120363. Epub 2022 Sep 24. PMID 36151975
- [Derived] Pandika D, Bailey JA, Oesterle S, Kuklinski MR. Young adult opioid misuse indicates a general tendency toward substance use and is strongly predicted by general substance use risk. Drug Alcohol Depend. 2022 Jun 1;235:109442. doi: 10.1016/j.drugalcdep.2022.109442. Epub 2022 Apr 6. PMID 35461085